CLINICAL TRIAL: NCT00003248
Title: A Randomized Phase II Study of Concurrent Fludarabine + Chimeric Anti-CD20 Monoclonal Antibody IDEC-C2B8 (Rituximab) [NSC# 687451] Induction Followed By Rituximab Consolidation In Untreated Patients With B-Cell Chronic Lymphocytic Leukemia
Brief Title: Fludarabine and Monoclonal Antibody Therapy in Treating Patients With Untreated B-cell Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9712; U10CA031946 (NIH); U01CA062475 (NIH); CLB-9712; CDR0000066128 (Registry Identifier: NCI Physicians Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-09-10 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia
Keywords: stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; fludarabine phosphate

ARMS (2):
- Arm I (Experimental): Patients receive fludarabine and chimeric anti-CD20 monoclonal antibody IDEC-C2B8 (rituximab) induction. Rituximab is administered IV over 4 hours on day 1, on day 3, and over 1 hour on day 5 of week 1. Subsequent doses are given over 1 hour on day 1 every 4 weeks for a total of 6 courses. Fludarabine IV is administered over 10-30 minutes daily for 5 days during weeks 1, 5, 9, 13, 17, and 21 for a total of 6 courses. Following the sixth course of fludarabine, patients undergo clinical staging and are then observed for an additional 2 months, after which they undergo repeat clinical staging, including bone marrow aspiration. Patients achieving a complete or partial response or stable disease then proceed to consolidation therapy consisting of weekly intravenous infusions of rituximab once weekly for 4 weeks.
  Patients are followed every 3 months for 1 year, and then every 6 months thereafter.
  Interventions: Biological: rituximab; Drug: fludarabine phosphate
- Arm II (Experimental): Patients receive fludarabine induction. Patients receive fludarabine IV over 10-30 minutes daily for 5 days during weeks 1, 5, 9, 13, 17, and 21 for a total of 6 courses. Patients then proceed as in arm I. Patients are followed every 3 months for 1 year, and then every 6 months thereafter.
  Interventions: Biological: rituximab; Drug: fludarabine phosphate

INTERVENTIONS:
Biological: rituximab
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining monoclonal antibody therapy with chemotherapy may kill more cancer cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of fludarabine given with or without monoclonal antibody therapy followed by monoclonal antibody therapy alone in treating patients who have untreated B-cell chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and toxicity profile of concurrent and consolidative chimeric anti-CD20 monoclonal antibody IDEC-C2B8 (rituximab) therapy compared to consolidative rituximab therapy in patients with chronic lymphocytic leukemia treated with fludarabine. II. Assess the complete response (CR) rate in patients receiving concurrent therapy with rituximab and fludarabine. III. Assess the frequency of conversion of a partial response (PR) to a CR or stable disease to either PR or CR in patients receiving consolidative therapy with rituximab. IV. Follow the effects of rituximab and fludarabine on the immunologic markers CD4, CD8, IgG, IgA, and IgM. V. Assess the progression-free and overall survival of these patients.

OUTLINE: This is a randomized study. Patients are stratified according to stage (I and II vs III and IV). Patients are assigned to 1 of 2 treatment arms. Arm I consists of fludarabine and chimeric anti-CD20 monoclonal antibody IDEC-C2B8 (rituximab) induction, and arm II consists of fludarabine induction. Arm I: Rituximab is administered IV over 4 hours on day 1, on day 3, and over 1 hour on day 5 of week 1. Subsequent doses are given over 1 hour on day 1 every 4 weeks for a total of 6 courses. Fludarabine IV is administered over 10-30 minutes daily for 5 days during weeks 1, 5, 9, 13, 17, and 21 for a total of 6 courses. Following the sixth course of fludarabine, patients undergo clinical staging and are then observed for an additional 2 months, after which they undergo repeat clinical staging, including bone marrow aspiration. Patients achieving a complete or partial response or stable disease then proceed to consolidation therapy consisting of weekly intravenous infusions of rituximab once weekly for 4 weeks. Arm II (Fludarabine Induction): Patients receive fludarabine IV over 10-30 minutes daily for 5 days during weeks 1, 5, 9, 13, 17, and 21 for a total of 6 courses. Patients then proceed as in arm I. Patients are followed every 3 months for 1 year, and then every 6 months thereafter.

PROJECTED ACCRUAL: A maximum of 100 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven B-cell chronic lymphocytic leukemia Stage I or II with evidence of active disease as defined by: Massive or progressive splenomegaly and/or lymphadenopathy Weight loss of greater than 10% within 6 months CALGB grade 2 or 3 fatigue Fevers of greater than 100.5 C or night sweats for over 2 weeks and no evidence of infection Progressive lymphocytosis Stage III or IV Patient registration on CALGB 9665 required

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: CALGB 0-3 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Creatinine no greater than 1.5 times upper limit of normal Other: No medical condition requiring chronic use of oral corticosteroids Direct antiglobulin test or direct Coombs test negative Not pregnant Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic: No prior biologic therapy for disease No concurrent erythropoietin Chemotherapy: No concurrent chemotherapy No prior chemotherapy for disease Endocrine: No concurrent chronic oral corticosteroids No prior corticosteroids for autoimmune complications developing since diagnosis No concurrent hormone therapy for disease related conditions No concurrent dexamethasone or other corticosteroid-based antiemetics Radiotherapy: No concurrent palliative radiotherapy Surgery: Not specified Other: No prophylactic therapy for viral, bacterial, or fungal infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 1998-03; Primary Completion 2003-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
progression-free survival | Up to 5 years
overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John C. Byrd, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (34):
- United States (34):
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Background] Morrison VA, Peterson BL, Rai KR, et al.: Alemtuzumab increases serious infections in patients with previously untreated chronic lymphocytic leukemia (CLL) receiving fludarabine-based therapy: a comparative analysis of 3 Cancer and Leukemia Group B studies (CALGB 9011, 9712, 19901). [Abstract] Blood 110 (11): A-756, 2007.
- [Background] Byrd JC, Rai K, Peterson BL, Appelbaum FR, Morrison VA, Kolitz JE, Shepherd L, Hines JD, Schiffer CA, Larson RA. Addition of rituximab to fludarabine may prolong progression-free survival and overall survival in patients with previously untreated chronic lymphocytic leukemia: an updated retrospective comparative analysis of CALGB 9712 and CALGB 9011. Blood. 2005 Jan 1;105(1):49-53. doi: 10.1182/blood-2004-03-0796. Epub 2004 May 11. PMID 15138165
- [Result] Woyach JA, Ruppert AS, Heerema NA, et al.: Treatment with fludarabine and rituximab produces extended overall survival (OS) and progression-free survival (PFS) in chronic lymphocytic leukemia (CLL) without increased risk of second malignancy: long-term follow up of CALGB study 9712. [Abstract] Blood 114 (22): A-539, 2009.
- [Result] Byrd JC, Gribben JG, Peterson BL, Grever MR, Lozanski G, Lucas DM, Lampson B, Larson RA, Caligiuri MA, Heerema NA. Select high-risk genetic features predict earlier progression following chemoimmunotherapy with fludarabine and rituximab in chronic lymphocytic leukemia: justification for risk-adapted therapy. J Clin Oncol. 2006 Jan 20;24(3):437-43. doi: 10.1200/JCO.2005.03.1021. Epub 2005 Dec 12. PMID 16344317
- [Result] Byrd JC, Peterson BL, Morrison VA, Park K, Jacobson R, Hoke E, Vardiman JW, Rai K, Schiffer CA, Larson RA. Randomized phase 2 study of fludarabine with concurrent versus sequential treatment with rituximab in symptomatic, untreated patients with B-cell chronic lymphocytic leukemia: results from Cancer and Leukemia Group B 9712 (CALGB 9712). Blood. 2003 Jan 1;101(1):6-14. doi: 10.1182/blood-2002-04-1258. Epub 2002 Jul 5. PMID 12393429
- [Result] Morrison VA, Byrd JC, Peterson BL, et al.: Adding Rituximab to Fludarabine therapy for patients with untreated chronic lymphocytic leukemia (CLL) does not Increase the risk of infection: Cancer and Leukemia Group B (CALGB) study 9712. [Abstract] Blood 102 (11 Pt 1): A-1606, 2003.
- [Result] Byrd JC, Peterson BL, Park K, et al.: Concurrent Rituximab and Fludarabine has a higher complete response rate than sequential treatment in untreated chronic lymphocytic leukemia (CLL) patients: results from CALGB 9712. [Abstract] Blood 98 (11 Pt 1): A-3212, 2001.
- [Result] Byrd JC, Peterson B, Park K, et al.: Rituximab added to Fludarabine improves response in previously untreated chronic lymphocytic leukemia: preliminary results from CALGB 9712. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-1116, 2001.